CLINICAL TRIAL: NCT07258914
Title: Feasibility and Efficacy of rTMS in Depression in Individuals With Autism Spectrum Disorder (ASD)
Brief Title: Feasibility and Efficacy of rTMS in Depression in Patients With Autism Spectrum Disorder (ASD)
Acronym: DEPASS'R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Center Guillaume Régnier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC24_01_CN_DEPASS'R; 2024-A01125-42 (Other: ANSM)
Record Dates: First submitted 2025-09-08; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Depression; Major Depressive Episode (MDE)
Keywords: Autism Spectrum Disorder; Depression; Major Depressive Episode (MDE); Transcranial Magnetic Stimulation; Repetitive Transcranial Magnectic Stimulation (rTMS); rTMS; Neurodivergent; executive and attentional function
MeSH Terms: conditions — Autism Spectrum Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASD patients with depression (Experimental): Patients receive 4 sessions of 10 minutes per day with a 50-minute interval between each session
  Interventions: Other: rTMS; Other: rTMS treatment with intermittent Theta Burst (ITBS)

INTERVENTIONS:
Other: rTMS — Patients receive 20 sessions of intermittent theta burst stimulation of the left CPFDL over 5 days (4 sessions of 10 minutes per day with a 50-minute interval between each session). The CPFDL is located using neuronavigation, which requires an MRI scan (without contrast agent injection) before the sessions.
Other: rTMS treatment with intermittent Theta Burst (ITBS) — rTMS (iTBS) treatment with stimulation of the left dorsolateral prefrontal cortex (DLPFC). Localization is performed using neuronavigation. There are four 10-minute sessions per day, with a 50-minute interval between each session.

SUMMARY:
Depression is a common complication of Autism Spectrum Disorder (ASD): it is four times more prevalent in people with ASD than in the general population.

However, treating depression in people with ASD is complicated by the lack of guidelines. Antidepressants appear to be less effective and less well tolerated than in the general population.

rTMS (repetitive transcranial magnetic stimulation) is a technique that stimulates the brain in a painless and non-invasive way. This technique is well tolerated and has very few side effects (headaches, fatigue). It is now used routinely in clinical practice to treat resistant depression, with satisfactory results.

A few studies using rTMS in depression in people with ASD have shown encouraging results and avenues for improvement.

It could therefore be interesting to conduct a therapeutic study with rTMS on depression in people with ASD, following the avenues for improvement proposed by previous studies.

The main objective is to evaluate the effectiveness of rTMS in depressed patients with ASD by looking at changes in mood before and after treatment. The investigator will also look at the effects on executive and attentional functions and repetitive behaviors, as well as treatment tolerance.

DETAILED DESCRIPTION:
Depression is a common comorbidity of autism spectrum disorder (ASD). Its prevalence is four times higher than in the neurotypical population, with specific symptoms, particularly irritability. However, the management of major depressive episodes (MDEs) in patients with ASD is complicated by the lack of specific recommendations for depression in ASD, while the effectiveness of pharmacological treatments is limited in this context.

rTMS (repetitive transcranial magnetic stimulation) is a technique that stimulates brain tissue in a non-invasive and painless manner, with good tolerance and few side effects. In the neurotypical population, it is used routinely in clinical practice to treat resistant EDMs, with satisfactory results.

To date, there are few studies on the treatment of depression in patients with ASD using TMS. Although these studies have certain limitations, they have shown encouraging results. These two studies are open-label studies involving fewer than 20 patients, but they show a significant improvement in depression scales before and after TMS treatment. The stimulation parameters (stimulation target: left dorsolateral prefrontal cortex, 15 to 30 sessions at a rate of one session per day, stimulation frequency of 10Hz for the first study and 50Hz in theta burst for the second) are those used in studies on depression in neurotypical depressed patients. In addition to the small sample size, these open-label studies have limitations in terms of parameter potentiation (target localisation, number of pulses per session and per day). It may therefore be worthwhile conducting a preliminary study to assess the feasibility and efficacy of rTMS in depressed ASD patients using an innovative accelerated, high-dose intermittent theta burst stimulation protocol with precise targeting of the stimulation site using neuronavigation and a detailed assessment of clinical depression in ASD, including irritability. Furthermore, an improvement in cognitive functions has been observed in neurotypical depressed patients receiving rTMS at the dorsolateral prefrontal cortex. It would therefore be interesting to study the impact of rTMS on executive and attentional functions using these innovative stimulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of ASD validated by a psychiatrist or line 2
* Patient aged 18 to 65...
* Patients suffering from EDM (MADRS greater than 20)
* No change in treatment in the month prior to inclusion
* Patients affiliated with or entitled to social security
* Patients who have received informed information about the study and have signed a consent form to participate in the study

Exclusion Criteria:

* Patients with psychiatric comorbidity (decompensated manic state, schizophrenic disorder)
* Pregnancy at the time of inclusion
* Patients with contraindications to rTMS and MRI (history of epilepsy, neurological stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid shunt, metal fragments in the eyes, claustrophobia)
* Adults under legal protection (legal guardianship, curatorship, trusteeship), persons deprived of their liberty, persons hospitalised under compulsion (SDT, SDRE).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Difference in MADRS (Montgomery-Asberg Depression Rating Scale ) score before versus after treatment. | From enrollment to the end of the data collecting process : 2 months.
  Upon inclusion, patients are assessed for mood using the MADRS.(inclusion criterion: MADRS>20).
  The primary endpoint is the change in MADRS score one week after the end of treatment and one month after the end of treatment.
  score ranges from 0 to 60. The higher the score, the more severe the disorder is.

SECONDARY OUTCOMES:
Assessment of changes in irritability before versus after treatment | from enrolment to one month after the end of the rTMS treatment
  Irritability is assessed with the Angst scale. A global score of 10 or more indicates irritability.
assessment of changes in attention functions | From enrolment to one week then 1 month after the end of the rTMS treatment
  Attentional functions are assessed using two subtests of the TAP (Test of Attentional Performance):
  * sustained attention : The test measures the ability to maintain attention over the long term with a high density of target stimuli.
  * Split Attention : The test explores the Ability to focus attention on two tasks simultaneously.
Evolution of any side effects | During the treatment, at each stimulation time
  Assessment of side effects of rTMS using the UKU scale
Assement of change in repetitive behaviors before versus after treatment | from enrolment and 1 month after the end of rTMS treatment
  BPI-1 (Behavior Problems Inventory) is an informant-based behaviour rating instrument that was designed to assess maladaptive behaviours in individuals with ASD. Its items fall into one of three sub-scales: Self-injurious Behavior (14 items), Stereotyped Behavior (24 items), and Aggressive/Destructive Behavior (11 items). Each item is rated on a frequency scale (0 = never to 4 = hourly), and a severity scale (0 = no problem to 3 = severe problem).
assessment of changes in mood aspects in terms of psychomotor decline before versus after rTMS treatment | from enrolment to one week then one month after the end of the rTMS treatment
  psychomotor decline is assessed with the depressive decline scale (ERD).This tool contains 14 items that describe the motor, verbal, ideational, hedonic, and cognitive behavior of depressed individuals. Each item is rated from 0 to 4 ( 1 expressing doubt about the pathological nature of the observed phenomenon).
assessment of changes in mood aspects in terms of depression before versus after rTMS treatment | From enrolment to one week then one month after the end of the rTMS treatment
  Depression is assessed with the Patient Health Questionnaire - 9 items (PHQ-9) This is a brief tool used to assess and measure the severity of depression. Items are rated on a scale from 0 to 3. The maximum score is 27 (major depression)
Assessment of changes in executive functions before versus after rTMS treatment | From enrolment and 1 month after the end of rTMS treatment
  The TMT (Trial Making Test) measures attention, visual screening ability, and processing speed. The Trail Making Test is scored by how long it takes to complete the test
Assessment of changes in executive functions before versus after rTMS treatment | From enrolment and 1 month after the end of rTMS treatment
  The Stroop test measures recognition reaction times to color stimuli, evaluating psychomotor speed and cognitive flexibility.
Assessment of changes in executive functions before versus after rTMS treatment | From enrolment and 1 month after the end of rTMS treatment
  The GO/NO GO task measures the ability to inhibit and the control of impulses

CONTACTS AND LOCATIONS:
Overall Officials: Cécilia NAUCZYCIEL, Doctor, Principal Investigator — Centre Hospitalier Guillaume Régnier
Locations (1):
- Centre Hospitalier Guillaume Régnier, Rennes, France

IPD SHARING:
Plan to Share IPD: No
Data about study protocol and clinical information will be available on request from other researchers.

REFERENCES:
- [Background] Smith JR, DiSalvo M, Green A, Ceranoglu TA, Anteraper SA, Croarkin P, Joshi G. Treatment Response of Transcranial Magnetic Stimulation in Intellectually Capable Youth and Young Adults with Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2023 Dec;33(4):834-855. doi: 10.1007/s11065-022-09564-1. Epub 2022 Sep 26. PMID 36161554
- [Background] Tong J, Zhang J, Jin Y, Liu W, Wang H, Huang Y, Shi D, Zhu M, Zhu N, Zhang T, Sun X. Impact of Repetitive Transcranial Magnetic Stimulation (rTMS) on Theory of Mind and Executive Function in Major Depressive Disorder and Its Correlation with Brain-Derived Neurotrophic Factor (BDNF): A Randomized, Double-Blind, Sham-Controlled Trial. Brain Sci. 2021 Jun 9;11(6):765. doi: 10.3390/brainsci11060765. PMID 34207545
- [Background] Noda Y, Fujii K, Mimura Y, Taniguchi K, Nakajima S, Kitahata R. A Case Series of Intermittent Theta Burst Stimulation Treatment for Depressive Symptoms in Individuals with Autistic Spectrum Disorder: Real World TMS Study in the Tokyo Metropolitan Area. J Pers Med. 2023 Jan 11;13(1):145. doi: 10.3390/jpm13010145. PMID 36675806
- [Background] Gwynette MF, Lowe DW, Henneberry EA, Sahlem GL, Wiley MG, Alsarraf H, Russo SB, Joseph JE, Summers PM, Lohnes L, George MS. Treatment of Adults with Autism and Major Depressive Disorder Using Transcranial Magnetic Stimulation: An Open Label Pilot Study. Autism Res. 2020 Mar;13(3):346-351. doi: 10.1002/aur.2266. Epub 2020 Jan 15. PMID 31944611
- [Background] Hudson CC, Hall L, Harkness KL. Prevalence of Depressive Disorders in Individuals with Autism Spectrum Disorder: a Meta-Analysis. J Abnorm Child Psychol. 2019 Jan;47(1):165-175. doi: 10.1007/s10802-018-0402-1. PMID 29497980